CLINICAL TRIAL: NCT05360888
Title: Comparative Effectiveness of Two Culturally-Centered Suicide Interventions for Alaska Native Youth
Brief Title: Suicide Intervention for Alaska Native Youth
Acronym: BeWeL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YY46Q97AEZA8
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Alaska Native Youth Aged 14 - 24; Suicide, Attempted; Suicidal Ideation; Alcohol Intoxication
Keywords: Alaska Native youth, suicide, prevention, culture
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation; Alcoholic Intoxication; Suicide

STUDY DESIGN:
Intervention Model Description: Half of the participants will be randomly assigned to Tools for Life, and the other half will receive Tools for Life plus a Motivational Interviewing Social Network intervention (MISN) and two booster sessions approximately 2 and 6 weeks post-intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tools for Life (Active Comparator): All youth will receive the Tools for Life (Qungasvik) intervention. Tools for Life is an evidence-based, community-developed intervention focused on providing protective cultural experiences for Alaska Native youth to address suicide risk and alcohol use.
  Interventions: Behavioral: Tools for Life
- Tools for Life + Motivational Interviewing Social Network intervention (MISN) (Active Comparator): Half of the youth will will also receive MISN in addition to the Tools for Life intervention. MISN is an evidence-based treatment that augments motivational interviewing with personal social network composition and structure visualization as a means to cultivating healthy social networks and cultural worlds.
  Interventions: Behavioral: Tools for Life + MISN

INTERVENTIONS:
Behavioral: Tools for Life — Tools for Life focuses on empowering youth to learn more about their culture and their identity.
  Arms: Tools for Life
Behavioral: Tools for Life + MISN — Tools for Life focuses on empowering youth to learn more about their culture and their identity. MISN focuses on helping youth get support from their community and social networks.
  Arms: Tools for Life + Motivational Interviewing Social Network intervention (MISN)

SUMMARY:
Two interventions will be delivered virtually to American Indian/Alaska Native youth who have been hospitalized with suicidal attempt, suicidal ideation, or associated risk behaviors, including alcohol-related injury.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial whereby Alaska Native (AN) youth who are hospitalized for suicide risk will be randomly assigned to either Qungasvik/Tools for Life or Tools for Life + Motivational Interviewing Social Network (MISN) intervention after their baseline survey, and followed up at 3-, 6-, and 12 months. All youth will receive Tools for Life and two 30-minute virtual follow-up visits (at 2- and 6-weeks post intervention) focused on connectivity to culture and obtaining support from intergenerational social networks in their home communities. Half of the youth will also receive MISN in addition to Tools for Life. Both interventions will be delivered virtually by a wellness team comprised of Alaska Native community behavioral health aides, prevention specialists and/or Elders who function in their communities as natural healers.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Alaska Native youth
* Between the ages of 14 and 24
* Admitted to the hospital for suicide attempt, ideation, or associated risk behaviors including alcohol-related injury or acute intoxication

Exclusion Criteria:

-

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Suicide intent/risk | Change from baseline to 3 months
  We will use the Suicidal Ideation Attributes Scale (SIDAS) [0 = Never, 10 = Always]
Suicide intent/risk | Change from baseline to 6 months
  We will use the Suicidal Ideation Attributes Scale (SIDAS) [0 = Never, 10 = Always]
Suicide intent/risk | Change from baseline to 12 months
  We will use the Suicidal Ideation Attributes Scale (SIDAS) [0 = Never, 10 = Always]
Depression | Change from baseline to 3 months
  Patient Health Questionnaire (PHQ-9) [0 -not at all to 3-nearly every day]
Depression | Change from baseline to 6 months
  Patient Health Questionnaire (PHQ-9) [0 -not at all to 3-nearly every day]
Depression | Change from baseline to 12 months
  Patient Health Questionnaire (PHQ-9) [0 -not at all to 3-nearly every day]
Anxiety | Change from baseline to 3 months
  Generalized Anxiety Disorder scale (GAD-7) [0 -not at all to 3-nearly every day]
Anxiety | Change from baseline to 6 months
  Generalized Anxiety Disorder scale (GAD-7) [0 -not at all to 3-nearly every day]
Anxiety | Change from baseline to 12 months
  Generalized Anxiety Disorder scale (GAD-7) [0 -not at all to 3-nearly every day]
Frequency of alcohol use | Change from baseline to 3 months
  Number of days used in the past 30 days. [ 0 to 30]
Frequency of alcohol use | Change from baseline to 6 months
  Number of days used in the past 30 days [ 0 to 30]
Frequency of alcohol use | Change from baseline to 12 months
  Number of days used in the past 30 days [ 0 to 30]
Alcohol use consequences | Change from baseline to 3 months
  Number of times in the past 3 months youth experience 4 different alcohol consequences [0 = Never to 6 = 20 or more times]
Alcohol use consequences | Change from baseline to 6 months
  Number of times in the past 3 months youth experience 4 different alcohol consequences [0 = Never to 6 = 20 or more times]
Alcohol use consequences | Change from baseline to 12 months
  Number of times in the past 3 months youth experience 4 different alcohol consequences [0 = Never to 6 = 20 or more times]

SECONDARY OUTCOMES:
Sobriety self-efficacy | Change from baseline to 3 months
  Three items ask how sure youth are about staying sober from alcohol from 1= def drink to 5 = def not drink
Sobriety self-efficacy | Change from baseline to 6 months
  Three items ask how sure youth are about staying sober from alcohol from 1= def drink to 5 = def not drink
Sobriety self-efficacy | Change from baseline to 12 months
  Three items ask how sure youth are about staying sober from alcohol from 1= def drink to 5 = def not drink
Intentions to be sober from alcohol | Change from baseline to 3 months
  Youth report on intentions to be sober in the next 6 months from 1 = def yes to 4 = def no
Intentions to be sober from alcohol | Change from baseline to 6 months
  Youth report on intentions to be sober in the next 6 months from 1 = def yes to 4 = def no
Intentions to be sober from alcohol | Change from baseline to 12 months
  Youth report on intentions to be sober in the next 6 months from 1 = def yes to 4 = def no
Social network composition | Change from baseline to 3 months
  Participants will be asked to name 15 contacts ("alters") who are at least 18 years of age. Participants will rate each of the 15 people on the same set of questions with categorical response options (about demographics, relationship quality, likelihood to use drugs, etc.). For each participant, the selected responses will be summed across all of the network alters and divided by 15 to produce network composition percentages of the whole set of alters named by the participant (% of AI/ANs, % who engage in heavy drinking).
Social network composition | Change from baseline to 6 months
  Participants will be asked to name 15 contacts ("alters") who are at least 18 years of age. Participants will rate each of the 15 people on the same set of questions with categorical response options (about demographics, relationship quality, likelihood to use drugs, etc.). For each participant, the selected responses will be summed across all of the network alters and divided by 15 to produce network composition percentages of the whole set of alters named by the participant (% of AI/ANs, % who engage in heavy drinking).
Social network composition | Change from baseline to 12 months
  Participants will be asked to name 15 contacts ("alters") who are at least 18 years of age. Participants will rate each of the 15 people on the same set of questions with categorical response options (about demographics, relationship quality, likelihood to use drugs, etc.). For each participant, the selected responses will be summed across all of the network alters and divided by 15 to produce network composition percentages of the whole set of alters named by the participant (% of AI/ANs, % who engage in heavy drinking).
Social network structure | Change from baseline to 3 months
  Participants will rate the relationship strength between each of the 15 named alters. For each alter pair participants will rate if the two people know each other and, if yes, have individuals connected recently. Measures of network structure (i.e., network "connectedness") will be constructed from the set of evaluations for each participant. For example, network "density" will be constructed for the network overall, which is calculated by summing the number of alter pairs who know each other and dividing by the total number of possible ties among 15 alters (105). Individual alter "centrality" will be calculated by summing the number of connections each individual alter has with other alters in the network.
Social network structure | Change from baseline to 6 months
  Participants will rate the relationship strength between each of the 15 named alters. For each alter pair participants will rate if the two people know each other and, if yes, have individuals connected recently. Measures of network structure (i.e., network "connectedness") will be constructed from the set of evaluations for each participant. For example, network "density" will be constructed for the network overall, which is calculated by summing the number of alter pairs who know each other and dividing by the total number of possible ties among 15 alters (105). Individual alter "centrality" will be calculated by summing the number of connections each individual alter has with other alters in the network.
Social network structure | Change from baseline to 12 months
  Participants will rate the relationship strength between each of the 15 named alters. For each alter pair participants will rate if the two people know each other and, if yes, have individuals connected recently. Measures of network structure (i.e., network "connectedness") will be constructed from the set of evaluations for each participant. For example, network "density" will be constructed for the network overall, which is calculated by summing the number of alter pairs who know each other and dividing by the total number of possible ties among 15 alters (105). Individual alter "centrality" will be calculated by summing the number of connections each individual alter has with other alters in the network.
Time spent around peers who use alcohol | Change from baseline to 3 months
  Participants will report on how much time is spent around peers who drink from 0 = never to 3 = often
Time spent around peers who use alcohol | Change from baseline to 6 months
  Participants will report on how much time is spent around peers who drink from 0 = never to 3 = often
Time spent around peers who use alcohol | Change from baseline to 12 months
  Participants will report on how much time is spent around peers who drink from 0 = never to 3 = often
Awareness of connectedness | Change from baseline to 3 months
  Youth report on feelings of connectedness to community, family and environment from 1 = strongly agree to 5 strongly disagree
Awareness of connectedness | Change from baseline to 6 months
  Youth report on feelings of connectedness to community, family and environment from 1 = strongly agree to 5 strongly disagree
Awareness of connectedness | Change from baseline to 12 months
  Youth report on feelings of connectedness to community, family and environment from 1 = strongly agree to 5 strongly disagree
Community protective factors | Change from baseline to 3 months
  Youth Community Protective Factors Scale. Youth report on feelings about different protective factors from 1 = strongly agree to 5 strongly disagree
Community protective factors | Change from baseline to 6 months
  Youth Community Protective Factors Scale Youth report on feelings about different community protective factors from 1 = strongly agree to 5 strongly disagree
Community protective factors | Change from baseline to 12 months
  Youth Community Protective Factors Scale Youth report on feelings about different community protective factors from 1 = strongly agree to 5 strongly disagree
Individual protective factors | Change from baseline to 3 months
  Youth report on feelings about different individual protective factors from 1 = strongly agree to 5 strongly disagree
Individual protective factors | Change from baseline to 6 months
  Youth report on feelings about different individual protective factors from 1 = strongly agree to 5 strongly disagree
Individual protective factors | Change from baseline to 12 months
  Youth report on feelings about different individual protective factors from 1 = strongly agree to 5 strongly disagree
Reasons for life | Change from baseline to 3 months
  Brief Reasons for Life Scale from 1 not at all important to 5 very important
Reasons for life | Change from baseline to 6 months
  Brief Reasons for Life Scale from 1 not at all important to 5 very important
Reasons for life | Change from baseline to 12 months
  Brief Reasons for Life Scale from 1 not at all important to 5 very important
Reflective processes | Change from baseline to 3 months
  The Reflective Processes scale taps a culturally patterned type of awareness and youth report from from 1 = strongly agree to 5 strongly disagree
Reflective processes | Change from baseline to 6 months
  The Reflective Processes scale taps a culturally patterned type of awareness and youth report from from 1 = strongly agree to 5 strongly disagree
Reflective processes | Change from baseline to 12 months
  The Reflective Processes scale taps a culturally patterned type of awareness and youth report from from 1 = strongly agree to 5 strongly disagree

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yukon-Kuskokwim Health Corporation, Bethel, Alaska
  - Tanana Chiefs Conference, Fairbanks, Alaska

IPD SHARING:
Plan to Share IPD: No
The investigators will share only deidentified, aggregate data.

REFERENCES:
- [Derived] Rasmus S, D'Amico EJ, Allen J, Nation C, John S, Joseph V, Rodriguez A, Alvarado G, Gittens AD, Palimaru AI, Brown RA, Kennedy DP, Woodward MJ, Parker J, McDonald K. A protocol for a randomized controlled comparative effectiveness trial of two brief interventions focused on social and cultural connectedness to reduce risk for suicide and substance misuse in young Alaska Native people. BMC Public Health. 2025 Oct 15;25(1):3503. doi: 10.1186/s12889-025-24710-z. PMID 41094443
- [Derived] Rasmus S, D'Amico EJ, Allen J, Nation C, John S, Joseph V, Rodriguez A, Alvarado G, Gittens AD, Palimaru AI, Brown RA, Kennedy DP, Woodward MJ, Parker J, McDonald K. Because We Love You (BeWeL): A protocol for a randomized controlled trial of two brief interventions focused on social and cultural connectedness to reduce risk for suicide and substance misuse in young Alaska Native people. Res Sq [Preprint]. 2024 Jan 22:rs.3.rs-3874293. doi: 10.21203/rs.3.rs-3874293/v1. PMID 38343833

DOCUMENTS (1):
  • Informed Consent Form (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT05360888/ICF_002.pdf